CLINICAL TRIAL: NCT02142829
Title: Pain Control in Bariatric Patients: A Prospective Trial Comparing the Effectiveness of EXPAREL(R) Versus the On-Q(R) Pain Ball
Brief Title: Pain Control in Bariatric Patients: EXPAREL(R) vs. the On-Q(R) Pain Ball
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: bariatric surgery, postoperative pain
MeSH Terms: conditions — Obesity; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL (Active Comparator): EXPAREL (bupivacaine liposome injectable suspension)
  Interventions: Drug: EXPAREL
- On-Q Pain Ball (Active Comparator): Device for delivering bupivacaine.
  Interventions: Drug: On-Q Pain Ball

INTERVENTIONS:
Drug: EXPAREL
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL
Drug: On-Q Pain Ball — bupivacaine HCl 0.25%
  Other Names: bupivacaine
  Arms: On-Q Pain Ball

SUMMARY:
This study was conducted to compare the effectiveness of two local pain control methods in bariatric patients by assessing the amount of postoperative pain and amount of postoperative pain medications needed. This information was used to determine which local anesthetic provided the best pain control.

DETAILED DESCRIPTION:
The investigators have previously utilized the On-Q® pain ball to obtain local control by continuous delivery of bupivacaine to pain fibers at the incision site. On-Q makes use of an implanted catheter and a continuous infusion pump that the patient carries with them typically for 48-72 hours after surgery. EXPAREL is a long-acting liposomal delivery vehicle that extends the life of bupivacaine in the surgical site for up to 72 hours. It can be injected in all trocar sites and offers another potential solution to patient pain control without the need for a catheter and the hardware needed to deliver the local anesthetic. Patient NRS (numerical rating scale) scores for postoperative pain and total medication consumed were used to assess the differences between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80, male or female

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) pain intensity scores | 4-6 hours postoperatively and in the mornings of postoperative Day 1 and Day 2
  The NRS was from 0 = no pain and 10 = worst pain.

SECONDARY OUTCOMES:
Postoperative opioid consumption | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Franchell Richard-Hamilton, MD, Principal Investigator — Bariatric Medical Institute of Texas
Locations (1):
- Bariatric Medical Institute of Texas, San Antonio, Texas, United States